CLINICAL TRIAL: NCT00798707
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of 2 Fixed Doses (25 and 50 mg/Day) of DVS SR Tablets in Adult Outpatients With Major Depressive Disorder
Brief Title: Study Evaluating Desvenlafaxine Succinate Sustained Release (DVS SR) in the Treatment of Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3151A1-3359; B2061003; 3151A1-3359-WW
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Results first posted 2011-06-06 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Desvenlafaxine succinate sustained-release 25 mg (Experimental)
  Interventions: Drug: Desvenlafaxine Succinate Sustained-Release (DVS SR)
- Desvenlafaxine succinate sustained-release 50 mg (Experimental)
  Interventions: Drug: Desvenlafaxine Succinate Sustained-Release (DVS SR)
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Desvenlafaxine Succinate Sustained-Release (DVS SR) — 25 mg tablet, once daily dosing for 8 weeks
  Arms: Desvenlafaxine succinate sustained-release 25 mg
Drug: Desvenlafaxine Succinate Sustained-Release (DVS SR) — 50 mg tablet, once daily dosing for 8 weeks
  Arms: Desvenlafaxine succinate sustained-release 50 mg
Drug: placebo — Matching placebo tablets (25 or 50 mg). Daily dosing for 10 +/- 4 days during a placebo lead-in period, and then 8 weeks during the double-blind period.
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to compare the antidepressant efficacy and safety of two doses of DVS SR (25 and 50 mg/day) in the treatment of adults with Major Depressive Disorder. The study will also assess changes in sexual function and general and functional quality of life outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult, outpatient with primary diagnosis of Major Depressive Disorder (depressive symptoms for at least 30 days prior to screening)
* Hamilton Psychiatric Rating Scale for Depression (HAM-D 17) total score of >= 20
* Clinical Global Impressions Scale-Severity (CGI-S) score of >= 4

Exclusion Criteria:

* Clinical instability - 25% or greater increase/decrease in HAM-D 17 total score from screening to baseline
* Significant risk of suicide as assessed by clinician judgement, HAM-D 17 and Columbia Suicide-Severity Rating Scale scores Other eligibility criteria also apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 709 (Actual)
Dates: Start 2008-12; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (63):
- United States (19):
  - Pfizer Investigational Site, Arcadia, California
  - Pfizer Investigational Site, Beverly Hills, California
  - Pfizer Investigational Site, Cerritos, California
  - Pfizer Investigational Site, Garden Grove, California
  - Pfizer Investigational Site, Los Alamitos, California
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Smyrna, Georgia
  - Pfizer Investigational Site, Libertyville, Illinois
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, East Providence, Rhode Island
  - Pfizer Investigational Site, Columbia, South Carolina
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Kirkland, Washington
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Brown Deer, Wisconsin
- Japan (44):
  - Pfizer Investigational Site, Nagoya, Aichi-ken
  - Pfizer Investigational Site, Toyoake, Aichi-ken
  - Pfizer Investigational Site, Noda, Chiba
  - Pfizer Investigational Site, Fukuoka, Fukuoka
  - Pfizer Investigational Site, Kitakyushu, Fukuoka
  - Pfizer Investigational Site, Fukushima, Fukushima
  - Pfizer Investigational Site, Shirakawa, Fukushima
  - Pfizer Investigational Site, Fujioka, Gunma
  - Pfizer Investigational Site, Kumagaya, Gunma
  - Pfizer Investigational Site, Hatsukaichi, Hiroshima
  - Pfizer Investigational Site, Hiroshima, Hiroshima
  - Pfizer Investigational Site, Kure, Hiroshima
  - Pfizer Investigational Site, Sapporo, Hokkaido
  - Pfizer Investigational Site, Kobe, Hyōgo
  - Pfizer Investigational Site, Kanazawa, Ishikawa-ken
  - Pfizer Investigational Site, Minamiashigara, Kanagawa
  - Pfizer Investigational Site, Yokohama, Kanagawa
  - Pfizer Investigational Site, Kumamoto, Kumamoto
  - Pfizer Investigational Site, Yatsushiro, Kumamoto
  - Pfizer Investigational Site, Kyoto, Kyoto
  - Pfizer Investigational Site, Matsumoto, Nagano
  - Pfizer Investigational Site, Osaka, Osaka
  - Pfizer Investigational Site, Sakai, Osaka
  - Pfizer Investigational Site, Kanzaka, Saga-ken
  - Pfizer Investigational Site, Misato, Saitama, Saitama
  - Pfizer Investigational Site, Saitama, Saitama
  - Pfizer Investigational Site, Kusatsu, Shiga
  - Pfizer Investigational Site, Bunkyo, Tokyo
  - Pfizer Investigational Site, Chiyoda City, Tokyo
  - Pfizer Investigational Site, Katsushika-ku, Tokyo
  - Pfizer Investigational Site, Kodaira, Tokyo
  - Pfizer Investigational Site, Minato, Tokyo
  - Pfizer Investigational Site, Nakano City, Tokyo
  - Pfizer Investigational Site, Setagaya City, Tokyo
  - Pfizer Investigational Site, Setagaya-ku, Tokyo
  - Pfizer Investigational Site, Shibuya City, Tokyo
  - Pfizer Investigational Site, Shinagawa, Tokyo
  - Pfizer Investigational Site, Shinjyuku, Tokyo
  - Pfizer Investigational Site, Suginami, Tokyo
  - Pfizer Investigational Site, tabashi City, Tokyo
  - Pfizer Investigational Site, Taitō City, Tokyo
  - Pfizer Investigational Site, Toshima City, Tokyo
  - Pfizer Investigational Site, Meguro City, Toyko
  - Pfizer Investigational Site, Ube, Yamaguchi

REFERENCES:
- [Derived] Zilcha-Mano S, Wang X, Wajsbrot DB, Boucher M, Fine SA, Rutherford BR. Trajectories of Function and Symptom Change in Desvenlafaxine Clinical Trials: Toward Personalized Treatment for Depression. J Clin Psychopharmacol. 2021 Sep-Oct 01;41(5):579-584. doi: 10.1097/JCP.0000000000001435. PMID 34183490
- [Derived] Soares CN, Zhang M, Boucher M. Categorical improvement in functional impairment in depressed patients treated with desvenlafaxine. CNS Spectr. 2019 Jun;24(3):322-332. doi: 10.1017/S1092852917000633. Epub 2017 Nov 15. PMID 29140227
- [Derived] McIntyre RS, Fayyad R, Mackell JA, Boucher M. Effect of metabolic syndrome and thyroid hormone on efficacy of desvenlafaxine 50 and 100 mg/d in major depressive disorder. Curr Med Res Opin. 2016;32(3):587-99. doi: 10.1185/03007995.2015.1136603. Epub 2016 Jan 13. PMID 26709542
- [Derived] McIntyre RS, Fayyad RS, Guico-Pabia CJ, Boucher M. A Post Hoc Analysis of the Effect of Weight on Efficacy in Depressed Patients Treated With Desvenlafaxine 50 mg/d and 100 mg/d. Prim Care Companion CNS Disord. 2015 Jun 4;17(3):10.4088/PCC.14m01741. doi: 10.4088/PCC.14m01741. eCollection 2015. PMID 26644956
- [Derived] Thase ME, Fayyad R, Cheng RF, Guico-Pabia CJ, Sporn J, Boucher M, Tourian KA. Effects of desvenlafaxine on blood pressure in patients treated for major depressive disorder: a pooled analysis. Curr Med Res Opin. 2015 Apr;31(4):809-20. doi: 10.1185/03007995.2015.1020365. Epub 2015 Mar 26. PMID 25758058
- [Derived] Iwata N, Tourian KA, Hwang E, Mele L, Vialet C. Efficacy and safety of desvenlafaxine 25 and 5050% shaded blockmg/day in a randomized, placebo-controlled study of depressed outpatients. J Psychiatr Pract. 2013 Jan;19(1):5-14. doi: 10.1097/01.pra.0000426323.59698.64. PMID 23334675
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3151A1-3359&StudyName=Study%20Evaluating%20Desvenlafaxine%20Succinate%20Sustained%20Release%20%28DVS%20SR%29%20in%20the%20Treatment%20of%20Major%20Depressive%20Disorder

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 907 potential participants were screened for this study. 813 participants were enrolled and received single-blind placebo during the screening period prior to randomization.
Groups:
- Placebo: Matching placebo tablets daily until Day 56 (Week 8) or early termination (ET) .
- DVS SR 25 mg: Desvenlafaxine Succinate Sustained Release (DVS SR) 25 mg daily until Day 56 (Week 8) or ET.
- DVS SR 50 mg: DVS SR 50 mg daily until Day 56 (Week 8) or ET.
Period: Overall Study
Arm/Group | Placebo | DVS SR 25 mg | DVS SR 50 mg
Started | 235 | 237 | 237
Treated | 231 | 232 | 236
Completed | 209 | 204 | 215
Not Completed | 26 | 33 | 22
Not completed — Adverse Event | 6 | 8 | 8
Not completed — Failed to return | 2 | 2 | 0
Not completed — Investigator | 0 | 1 | 2
Not completed — Lack of Efficacy | 2 | 2 | 1
Not completed — Lost to Follow-up | 5 | 6 | 6
Not completed — Other | 0 | 1 | 0
Not completed — Protocol Violation | 4 | 0 | 2
Not completed — Withdrawal by Subject | 3 | 8 | 2
Not completed — Randomized not treated | 4 | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | DVS SR 25 mg | DVS SR 50 mg | Total
Number analyzed (Participants) | 231 | 232 | 236 | 699
Age Continuous [Mean (Standard Deviation); unit: Years] | 40.26 (12.32) | 40.19 (11.88) | 38.59 (12.08) | 39.67 (12.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 127 | 131 | 386
  Male | 103 | 105 | 105 | 313
Hamilton Psychiatric Scale for Depression-17 item (HAM-D17) total score [Mean (Standard Deviation); unit: Units on a scale] — HAM-D17: a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression. Items are scored on either a 3 point (0 to 2) or a 5 point scale (0 to 4), with 0=none/absent and 4=most severe, for a maximum total score of 50.
  Units on a scale | 23.06 (2.59) | 23.08 (2.93) | 22.81 (2.61) | 22.98 (2.71)
Clinical Global Impressions Scale-Severity of Illness (CGI-S) Score [Mean (Standard Deviation); unit: Units on a scale] — CGI-S: 7-point clinician rated scale to assess severity of participant's current illness state; range: 1 (normal - not ill at all) to 7 (among the most extremely ill patients). Higher score = more affected.
  Units on a scale | 4.39 (0.59) | 4.35 (0.57) | 4.33 (0.56) | 4.36 (0.58)
Montgomery-Asberg Depression Rating Scale (MADRS) total score [Mean (Standard Deviation); unit: Units on a scale] — MADRS measures the overall severity of depressive symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
  Units on a scale | 28.19 (5.74) | 28.08 (5.46) | 28.21 (5.38) | 28.16 (5.52)
HAM-D6 total score [Mean (Standard Deviation); unit: Units on a scale] — HAM-D6: a standardized, clinician-administered rating scale that assesses 6 items associated with major depression and is a subset of the HAM-D17. HAM-D6 score ranges from 0-22. The scale uses HAM-D17 items: 1, 2, 7, 8, 10 and 13. Item 13 is scored 0-2 and all others are scored 0-4.
  Units on a scale | 12.58 (1.79) | 12.61 (1.77) | 12.43 (1.75) | 12.54 (1.77)
Sheehan Disability Scale (SDS) Total Score [Mean (Standard Deviation); unit: Units on a scale] — SDS: a self-administered tool that measures functional impairment in 3 domains: Work/School, Social Life, and Family Life/Home Responsibilities.Participant rates extent to which each of these domains are impaired by his/her symptoms using 10 point visual analog scale:(0=not at all impaired,10=extremely impaired) for total maximum score of 30.
  Units on a scale | 16.31 (7.78) | 17.02 (7.34) | 16.39 (7.27) | 16.57 (7.46)
World Health Organization 5-Item Well-Being Index (WHO-5) [Mean (Standard Deviation); unit: Units on a scale] — WHO-5 evaluates positive psychological well-being. WHO-5 consists of 5 questions and each is rated on a 6-point scale. The total score ranges from 0 to 25 ( 0= worst possible quality of life; 25=best possible quality of life).
  Units on a scale | 7.21 (4.47) | 6.89 (3.99) | 7.18 (4.34) | 7.09 (4.27)
Participants with Sexual dysfunction [Number; unit: Percentage of Participants] — Arizona Sexual Experiences Scale (ASEX) includes 5 questions that evaluate sexual function exclusively during week prior to completion in the following areas: libido, excitability and ability to reach orgasm. Sexual dysfunction=ASEX total score of 19 or greater, or a score of 5 or greater on any item, or a score of 4 or greater on any 3 items.
  Percentage of Participants | 66.4 | 66.1 | 62.3 | 194.8
Participants with Columbia Suicide-Severity Rating Scale (C-SSRS) total score [Number; unit: Participants] — C-SSRS was mapped into Columbia Classification Algorithm of Suicide Assessment (C-CASA)(1-4) to prospectively assess whether participants experienced: completed suicide(1),suicide attempt(2),preparatory acts toward imminent suicidal behavior(3),suicidal ideation,any suicidal behavior and ideation(4).Participants with "yes" response were reported.
  Participants
    Completed Suicide | 0 | 0 | 0 | 0
    Suicide attempt | 0 | 0 | 0 | 0
    Preparatory acts toward imminent suicidal behavior | 0 | 0 | 0 | 0
    Suicidal ideation | 31 | 45 | 37 | 113

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HAM-D17 Total Score at the Final On-therapy (FOT)Evaluation (Week 8 or ET)
Description: HAM-D17: a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression. Items are scored on either a 3 point (0 to 2) or a 5 point scale (0 to 4), with 0=none/absent and 4=most severe, for a maximum total score of 50.
Time Frame: Baseline and Week 8 (or ET)
Population: Intent-To-Treat (ITT) Population:all randomly assigned participants with baseline primary efficacy evaluation, had taken at least 1 dose of double-blind drug and 1 primary efficacy evaluation after first dose of double-blind drug. If participant had missing value at any visit, last observation carried forward (LOCF) method of imputation was used.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | DVS SR 25 mg | DVS SR 50 mg
Number analyzed (Participants) | 231 | 232 | 236
Units on a scale | -8.52 (0.44) | -8.98 (0.44) | -10.02 (0.44)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 25 mg; An analysis of covariance (ANCOVA) model with treatment and as a factor and the baseline HAM-D17 total score as a covariate was used to compare each DVS SR dose to placebo. The comparison was performed at the 0.05 level overall; Test type: Superiority or Other; p = 0.452, ANCOVA — A Hochberg step-up procedure was used to control for the multiplicity associated with multiple active dose arms; Mean Difference (Final Values) = 0.47, 95% CI 2-sided [-0.75 to 1.69]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.016, ANCOVA — A Hochberg step-up procedure was used to control for the multiplicity associated with multiple active dose arms; Mean Difference (Final Values) = 1.50, 95% CI 2-sided [0.28 to 2.72]

2. Secondary Outcome: Number of Participants With Categorical Scores on CGI-Improvement (CGI-I) at FOT Evaluation (Week 8 or ET)
Description: CGI-I: 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Higher score = more affected.
Time Frame: Week 8 (or ET)
Population: ITT Population included all randomly assigned participants who had baseline primary efficacy evaluation, had taken at least 1 dose of double-blind study drug, and had at least 1 primary efficacy evaluation after first dose of double-blind study drug. If participant had a missing value at any visit, LOCF method of imputation was used.
Measure: Number; unit: Participants
Arm/Group | Placebo | DVS SR 25 mg | DVS SR 50 mg
Number analyzed (Participants) | 231 | 232 | 236
Participants
  1=Very much improved | 48 | 57 | 68
  2=Much improved | 61 | 61 | 62
  3=Minimally improved | 62 | 70 | 61
  4=No change | 52 | 37 | 36
  5=Minimally worse | 4 | 5 | 4
  6=Much worse | 3 | 1 | 5
  7=Very much worse | 1 | 1 | 0
Statistical Analysis 1: Comparison: Placebo vs DVS SR 25 mg; Each DVS SR dose was separately compared to placebo. To control the study-wise type I error rate across the primary and the key secondary endpoints, as well as across the 2 active dose arms, testing of the key secondary hypothesis occurred only when both active doses were superior to placebo on the primary endpoint; Test type: Superiority or Other; p = 0.160, Cochran-Mantel-Haenszel — In this case, multiplicity arising from testing key secondary hypotheses in both doses was controlled by a Hochberg step-up procedure. p-Value obtained for the alternative hypothesis of 'Row mean scores differences'
Statistical Analysis 2: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.028, Cochran-Mantel-Haenszel — In this case, multiplicity arising from testing key secondary hypotheses in both doses was controlled by a Hochberg step-up procedure.p-Value obtained for the alternative hypothesis of 'Row mean scores differences'

3. Secondary Outcome: Change From Baseline in Mean CGI-S Score at FOT Evaluation (Week 8 or ET)
Description: CGI-S: 7-point clinician rated scale to assess severity of participant's current illness state; range: 1 (normal - not ill at all) to 7 (among the most extremely ill patients). Higher score = more affected.
Time Frame: Baseline and Week 8 (or ET)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | DVS SR 25 mg | DVS SR 50 mg
Number analyzed (Participants) | 231 | 232 | 236
Units on a scale | -1.03 (0.07) | -1.22 (0.07) | -1.24 (0.07)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 25 mg; Analysis was conducted using ANCOVA on the change from baseline with treatment as a factor and corresponding baseline value as a covariate; Test type: Superiority or Other; p = 0.066, ANCOVA; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.01 to 0.39]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.038, ANCOVA; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [0.01 to 0.41]

4. Secondary Outcome: Change From Baseline in MADRS Total Score at FOT Evaluation (Week 8 or ET)
Description: MADRS measures the overall severity of depressive symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
Time Frame: Baseline and Week 8 (or ET)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | DVS SR 25 mg | DVS SR 50 mg
Number analyzed (Participants) | 229 | 231 | 235
Units on a scale | -9.23 (0.61) | -10.23 (0.60) | -11.29 (0.60)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 25 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.242, ANCOVA; Mean Difference (Final Values) = 1.00, 95% CI 2-sided [-0.68 to 2.68]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.016, ANCOVA; Mean Difference (Final Values) = 2.06, 95% CI 2-sided [0.39 to 3.73]

5. Secondary Outcome: Change From Baseline in HAM-D6 Total Score at FOT Evaluation (Week 8 or ET)
Description: HAM-D6: a standardized, clinician-administered rating scale that assesses 6 items characteristically associated with major depression and is a subset of HAM-D17. HAM-D6 score ranges from 0-22. The scale uses HAM-D17 items: 1, 2, 7, 8, 10 and 13. Item 13 is scored 0-2 and all others are scored 0-4.
Time Frame: Baseline and Week 8 (or ET)
Population: ITT Population: all randomly assigned participants with baseline primary efficacy evaluation had taken at least 1 dose of double-blind drug and 1 primary efficacy evaluation after first dose of double-blind drug. If participant had missing value at any visit,LOCF method of imputation was used.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | DVS SR 25 mg | DVS SR 50 mg
Number analyzed (Participants) | 231 | 232 | 236
Units on a scale | -4.94 (0.26) | -5.03 (0.26) | -5.65 (0.25)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 25 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.802, ANCOVA; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.62 to 0.80]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.048, ANCOVA; Median Difference (Final Values) = 0.72, 95% CI 2-sided [0.01 to 1.43]

6. Secondary Outcome: Number of Participants With a Response on the HAM-D17 at FOT Evaluation (Week 8 or ET)
Description: A HAM-D17 responder was defined as a participant with a 50% or greater decrease from baseline in HAM-D17 score. HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression. Individual items are scored on either a 3 point (0 to 2) or a 5 point scale (0 to 4), with 0=none/absent and 4=most severe, for a maximum total score of 50.
Time Frame: Week 8 (or ET)
Population: ITT Population: all randomly assigned participants with baseline primary efficacy evaluation had taken at least 1 dose of double-blind drug and 1 primary efficacy evaluation after first dose of double-blind drug. If participant had missing value at any visit, LOCF method of imputation was used.
Measure: Number; unit: Participants
Arm/Group | Placebo | DVS SR 25 mg | DVS SR 50 mg
Number analyzed (Participants) | 231 | 232 | 236
Participants | 80 | 97 | 109
Statistical Analysis 1: Comparison: Placebo vs DVS SR 25 mg; Analysis was conducted using a logistic regression model with treatment as a factor and baseline HAM-D17 score as a covariate; Test type: Superiority or Other; p = 0.1099, Regression, Logistic; Odds Ratio (OR) = 1.363, 95% CI 2-sided [0.93 to 1.99]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.0154, Regression, Logistic; Odds Ratio (OR) = 1.591, 95% CI 2-sided [1.09 to 2.32]

7. Secondary Outcome: Number of Participants in Remission Based on the HAM-D17 at FOT Evaluation (Week 8 or ET)
Description: Remission was defined as a HAM-D17 score of less than or equal to 7. HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression. Individual items are scored on either a 3 point (0 to 2) or a 5 point scale (0 to 4), with 0=none/absent and 4=most severe, for a maximum total score of 50.
Time Frame: Week 8 (or ET)
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Placebo | DVS SR 25 mg | DVS SR 50 mg
Number analyzed (Participants) | 231 | 232 | 236
Participants | 44 | 40 | 62
Statistical Analysis 1: Comparison: Placebo vs DVS SR 25 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.5929, Regression, Logistic; Odds Ratio (OR) = 0.878, 95% CI 2-sided [0.54 to 1.41]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.0852, Regression, Logistic; Odds Ratio (OR) = 1.474, 95% CI 2-sided [0.95 to 2.29]

8. Secondary Outcome: Number of Participants With a Response on the MADRS Score at FOT Evaluation (Week 8 or ET)
Description: A MADRS responder was defined as a participant with a 50% or greater decrease from baseline in MADRS score. It measures the overall severity of depressive symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
Time Frame: Week 8 (or ET)
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Placebo | DVS SR 25 mg | DVS SR 50 mg
Number analyzed (Participants) | 229 | 231 | 235
Participants | 68 | 81 | 102
Statistical Analysis 1: Comparison: Placebo vs DVS SR 25 mg; Analysis was conducted with a logistic regression model with treatment as a factor and baseline MADRS score as a covariate; Test type: Superiority or Other; p = 0.2232, Regression, Logistic; Odds Ratio (OR) = 1.277, 95% CI 2-sided [0.86 to 1.89]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.0022, Regression, Logistic; Odds Ratio (OR) = 1.827, 95% CI 2-sided [1.24 to 2.69]

9. Secondary Outcome: Number of Participants With a Response on the CGI-I Score at FOT Evaluation (Week 8 or ET)
Description: CGI-I responder was defined as a participant with a score of 1 (very much improved) or 2 (much improved) on the CGI-I. CGI-I: 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Higher score = more affected.
Time Frame: Week 8 (or ET)
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Placebo | DVS SR 25 mg | DVS SR 50 mg
Number analyzed (Participants) | 231 | 232 | 236
Participants | 109 | 118 | 130
Statistical Analysis 1: Comparison: Placebo vs DVS SR 25 mg; Analysis was conducted with a logistic regression model with treatment as a factor; Test type: Superiority or Other; p = 0.4313, Regression, Logistic; Odds Ratio (OR) = 1.158, 95% CI 2-sided [0.80 to 1.67]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 50 mg; Analysis was conducted with a logistic regression model with treatment as a factor; Test type: Superiority or Other; p = 0.0888, Regression, Logistic; Odds Ratio (OR) = 1.372, 95% CI 2-sided [0.95 to 1.97]

10. Other Pre Specified Outcome: Population Pharmacokinetics for Desvenlafaxine Plasma Concentrations
Description: Relationship of demographic variables (age, gender, food, race, creatinine, aspartate aminotransaminase, alanine transaminase, bilirubin and concomitant medications) were examined by fitting measured DVS plasma concentrations to a 1 compartment model with first order absorption. Demographic variables were examined for clearance (CL/F), volume of distribution (V/F), Steady Area under Curve (AUC) using nonlinear mixed effects modeling. Final parameter estimates for demographic factors effecting CL/F, V/F and AUC were determined.
Time Frame: Week 2, 4 and 8 (or ET)
Population: PK population; data was insufficient examine the effect of demographic variables on the PK of desvenlafaxine. Parameter values were calculated for variables altering CL/F, AUC and V/F. Population parameters from nonlinear mixed effects modeling were not summarized as descriptive statistics.
Measure: Mean (Standard Deviation); unit: nanogram(ng)/mL
Arm/Group | Placebo | DVS SR 25 mg | DVS SR 50 mg
Number analyzed (Participants) | 0 | 0 | 0

11. Other Pre Specified Outcome: Change From Baseline in SDS at FOT Evaluation (Week 8 or ET)
Description: SDS: a self-administered tool that measures functional impairment in 3 domains: Work/School, Social Life, and Family Life/Home Responsibilities. The participant rates the extent to which each of these domains is impaired by his/her symptoms using a 10 point visual analog scale: (0=not at all impaired, 10=extremely impaired) for a total maximum score of 30.
Time Frame: Baseline and Week 8 (or ET)
Population: ITT Population included all randomly assigned participants who had baseline primary efficacy evaluation,had taken at least 1 dose of double-blind study drug,had at least 1 primary efficacy evaluation after first dose of double-blind drug.'n' is participants who received drug and were evaluated for measure at timepoint for each group respectively.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | DVS SR 25 mg | DVS SR 50 mg
Number analyzed (Participants) | 231 | 232 | 236
Units on a scale
  Total Score (n=227,224,235) | -2.17 (0.43) | -3.26 (0.43) | -3.23 (0.42)
  Work/Studies Component (n=227,225,235) | -0.77 (0.16) | -1.07 (0.15) | -1.12 (0.15)
  Social Life Component (n=229,231,235) | -0.86 (0.16) | -1.26 (0.15) | -1.21 (0.15)
  Family Life/Home Responsibilities (n=14,2,13) | -0.54 (0.88) | -1.83 (2.12) | -0.97 (0.89)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 25 mg; Analysis was conducted using ANCOVA on the change from baseline with treatment as a factor and corresponding baseline value as a covariate for total score; Test type: Superiority or Other; p = 0.073, ANCOVA; Mean Difference (Final Values) = 1.09, 95% CI 2-sided [-0.10 to 2.29]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.078, ANCOVA; Median Difference (Final Values) = 1.06, 95% CI 2-sided [-0.12 to 2.24]
Statistical Analysis 3: Comparison: Placebo vs DVS SR 25 mg; Analysis was conducted using ANCOVA on the change from baseline with treatment as a factor and corresponding baseline value as a covariate for work/studies component score; Test type: Superiority or Other; p = 0.176, ANCOVA; Mean Difference (Final Values) = 0.30, 95% CI 2-sided [-0.13 to 0.73]
Statistical Analysis 4: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 11, analysis 3]; Test type: Superiority or Other; p = 0.109, ANCOVA; Mean Difference (Final Values) = 0.35, 95% CI 2-sided [-0.08 to 0.77]
Statistical Analysis 5: Comparison: Placebo vs DVS SR 25 mg; Analysis was conducted using ANCOVA on the change from baseline with treatment as a factor and corresponding baseline value as a covariate for social life component score; Test type: Superiority or Other; p = 0.064, ANCOVA; Mean Difference (Final Values) = 0.41, 95% CI 2-sided [-0.02 to 0.84]
Statistical Analysis 6: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 11, analysis 5]; Test type: Superiority or Other; p = 0.104, ANCOVA; Mean Difference (Final Values) = 0.35, 95% CI 2-sided [-0.07 to 0.78]
Statistical Analysis 7: Comparison: Placebo vs DVS SR 25 mg; Analysis was conducted using ANCOVA on the change from baseline with treatment as a factor and corresponding baseline value as a covariate for family life/home responsibilities component score; Test type: Superiority or Other; p = 0.538, ANCOVA; Mean Difference (Final Values) = 1.29, 95% CI 2-sided [-2.98 to 5.57]
Statistical Analysis 8: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 11, analysis 7]; Test type: Superiority or Other; p = 0.689, ANCOVA; Mean Difference (Final Values) = 0.43, 95% CI 2-sided [-1.76 to 2.62]

12. Other Pre Specified Outcome: Change From Baseline in WHO-5 Total Score at FOT Evaluation (Week 8 or ET)
Description: WHO-5 evaluates positive psychological well-being. WHO-5 consists of 5 questions and each is rated on a 6-point scale. The total score ranges from 0 to 25 (0= worst possible quality of life; 25=best possible quality of life).
Time Frame: Baseline and Week 8 (or ET)
Population: as for outcome 6
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | DVS SR 25 mg | DVS SR 50 mg
Number analyzed (Participants) | 229 | 231 | 235
Units on a scale | 2.62 (0.31) | 3.43 (0.31) | 3.25 (0.31)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 25 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.066, ANCOVA; Mean Difference (Final Values) = -0.81, 95% CI 2-sided [-1.67 to 0.05]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.150, ANCOVA; Mean Difference (Final Values) = -0.63, 95% CI 2-sided [-1.48 to 0.23]

13. Other Pre Specified Outcome: Percentage of Participants With Sexual Dysfunction at FOT Evaluation (Week 8 or ET)
Description: ASEX scale includes 5 questions that evaluate sexual function exclusively during the week prior to completion in the following areas: libido, excitability and ability to reach orgasm. Sexual dysfunction=an ASEX total score of 19 or greater, or a score of 5 or greater on any item, or a score of 4 or greater on any 3 items. Participants who have had no sexual activity during the prior week should be instructed to not complete questions 3 through 5.
Time Frame: Week 8 (or ET)
Population: The safety population included all participants randomly assigned to treatment who had taken at least 1 dose of double-blind study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | DVS SR 25 mg | DVS SR 50 mg
Number analyzed (Participants) | 109 | 112 | 113
Percentage of Participants | 55.0 | 52.7 | 55.8
Statistical Analysis 1: Comparison: Placebo vs DVS SR 25 mg; Analysis was conducted using a logistic regression model with treatment and gender as factors and baseline sexual dysfunction status as a covariate; Test type: Superiority or Other; p = 0.8758, Regression, Logistic; Odds Ratio (OR) = 0.951, 95% CI 2-sided [0.51 to 1.78]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.6397, Regression, Logistic; Odds Ratio (OR) = 1.165, 95% CI 2-sided [0.61 to 2.21]

14. Other Pre Specified Outcome: Number of Participants With Categorical Scores on the C-SSRS at FOT Evaluation (Week 8 or ET)
Description: C-SSRS mapped into C-CASA(1-7) to assess whether participant:completed suicide(1),suicide attempt(2)(response of "Yes" on "Actual Attempt"),preparatory acts toward imminent suicidal behavior (3)("Yes" on "Preparatory Acts or Behavior"),suicidal ideation (4)("Yes" on "Wish to be dead","Non-Specific Active Suicidal Thoughts","Active Suicidal Ideation with methods without Intent to Act or Some Intent to Act,without Specific Plan or with Specific Plan and Intent),any suicidal behavior or ideation,self-injurious behaviour(7)("Yes" on "Has subject engaged in Non-suicidal Self-Injurious Behavior").
Time Frame: Week 8 (or ET)
Population: as for outcome 13
Measure: Number; unit: Participants
Arm/Group | Placebo | DVS SR 25 mg | DVS SR 50 mg
Number analyzed (Participants) | 231 | 232 | 236
Participants
  Completed suicide | 0 | 0 | 0
  Suicide attempt | 0 | 0 | 1
  Preparatory acts toward imminent suicidal behavior | 0 | 0 | 0
  Suicidal ideation | 42 | 50 | 47
  Any suicidal behavior and/or ideation | 42 | 50 | 47
  Self-injurious behavior, no suicidal intent | 0 | 1 | 1

15. Other Pre Specified Outcome: Discontinuation-Emergent Signs and Symptoms (DESS) Total Score
Description: DESS: a clinician-administered 43-item assessment that evaluates discontinuation-emergent symptoms resulting from the withdrawal from test article. The DESS total score is the sum of the number of "new symptoms" and "old (but worse) symptoms" (1) and 0 for "old and unchanged symptom," "absent," or "old symptom but improved" for a total possible range of 0 to 43. A higher score indicates more symptoms.
Time Frame: Week 8 to 10 (or ET)
Population: Analysis included completers for exposure (those whose exposure duration was at least 53 days) among safety population. 'n' is participants who received drug and were evaluated for measure at timepoint for each group respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | DVS SR 25 mg | DVS SR 50 mg
Number analyzed (Participants) | 231 | 232 | 236
Units on a scale
  Week 8 (or ET) (n=96,88,100) | 0.67 (1.62) | 0.63 (1.30) | 0.62 (1.53)
  Week 9 (or ET + 1 week) (n=93,84,98) | 1.08 (2.68) | 1.38 (2.58) | 1.50 (2.81)
  Week 10 (or ET + 2 weeks) (n=83,76,89) | 0.94 (2.28) | 0.74 (1.23) | 0.63 (1.60)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 25 mg; To address the multiplicity effect inherent in these comparisons, adjusted p-values based on the false discovery rate were used at Week 8 (or ET); Test type: Superiority or Other; p = 0.847, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p = 0.847, t-test, 2 sided
Statistical Analysis 3: Comparison: Placebo vs DVS SR 25 mg; To address the multiplicity effect inherent in these comparisons, adjusted p-values based on the false discovery rate were used at Week 9 (or ET + 1 week); Test type: Superiority or Other; p = 0.720, t-test, 2 sided
Statistical Analysis 4: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 15, analysis 3]; Test type: Superiority or Other; p = 0.720, t-test, 2 sided
Statistical Analysis 5: Comparison: Placebo vs DVS SR 25 mg; To address the multiplicity effect inherent in these comparisons, adjusted p-values based on the false discovery rate were used at Week 10 (or ET + 2 weeks); Test type: Superiority or Other; p = 0.720, t-test, 2 sided
Statistical Analysis 6: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p = 0.720, t-test, 2 sided

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | DVS SR 25 mg | DVS SR 50 mg
Serious Adverse Events (participants affected / at risk) | 3/231 | 1/232 | 5/236
Other Adverse Events (participants affected / at risk) | 158/231 | 160/232 | 174/236
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=231) | DVS SR 25 mg (N=232) | DVS SR 50 mg (N=236)
Chest discomfort (General disorders) | 0 | 0 | 1
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pancreatic neuroendocrine tumour metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Grand mal convulsion (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 2
Hallucination, auditory (Psychiatric disorders) | 0 | 0 | 1
Homicidal ideation (Psychiatric disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=231) | DVS SR 25 mg (N=232) | DVS SR 50 mg (N=236)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 3 | 4 | 2
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Hyperacusis (Ear and labyrinth disorders) | 2 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 6 | 1 | 3
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 4
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1
Hyperprolactinaemia (Endocrine disorders) | 1 | 0 | 0
Abnormal sensation in eye (Eye disorders) | 0 | 1 | 0
Accommodation disorder (Eye disorders) | 0 | 0 | 1
Asthenopia (Eye disorders) | 0 | 1 | 0
Blepharospasm (Eye disorders) | 2 | 0 | 0
Corneal disorder (Eye disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 1 | 1 | 2
Eye pain (Eye disorders) | 0 | 1 | 3
Eye swelling (Eye disorders) | 0 | 1 | 0
Foreign body sensation in eyes (Eye disorders) | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 1
Scintillating scotoma (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 5 | 7
Visual impairment (Eye disorders) | 0 | 1 | 0
Vitreous detachment (Eye disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 3 | 1 | 7
Abdominal distension (Gastrointestinal disorders) | 3 | 4 | 2
Abdominal mass (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 4
Abdominal pain upper (Gastrointestinal disorders) | 7 | 5 | 8
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 4 | 6 | 13
Diarrhoea (Gastrointestinal disorders) | 14 | 15 | 14
Dry mouth (Gastrointestinal disorders) | 10 | 15 | 10
Dyspepsia (Gastrointestinal disorders) | 6 | 4 | 6
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 2 | 2 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0
Glossitis (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 15 | 23 | 36
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 2 | 2
Tongue disorder (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 4 | 1
Vomiting (Gastrointestinal disorders) | 7 | 5 | 7
Asthenia (General disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 2 | 1 | 1
Chills (General disorders) | 2 | 1 | 1
Energy increased (General disorders) | 1 | 0 | 0
Facial pain (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 5 | 5 | 11
Feeling abnormal (General disorders) | 0 | 1 | 1
Feeling cold (General disorders) | 0 | 0 | 1
Feeling jittery (General disorders) | 0 | 0 | 2
Gait disturbance (General disorders) | 1 | 0 | 2
Hangover (General disorders) | 0 | 0 | 1
Hunger (General disorders) | 0 | 1 | 0
Irritability (General disorders) | 3 | 7 | 6
Loss of control of legs (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 2 | 2 | 0
Mass (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Oedema (General disorders) | 0 | 2 | 0
Oedema peripheral (General disorders) | 1 | 1 | 0
Pain (General disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 4 | 1 | 1
Sluggishness (General disorders) | 1 | 0 | 0
Thirst (General disorders) | 3 | 3 | 7
Vessel puncture site haematoma (General disorders) | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1 | 3
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 1 | 0
Abscess jaw (Infections and infestations) | 0 | 0 | 1
Acne pustular (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0
Conjunctivitis infective (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 1 | 1
Enteritis infectious (Infections and infestations) | 0 | 1 | 0
Gastritis viral (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 3 | 2 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
H1N1 influenza (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Hordeolum (Infections and infestations) | 1 | 1 | 0
Infected bites (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 5 | 4
Laryngitis (Infections and infestations) | 0 | 1 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 37 | 26 | 30
Oral herpes (Infections and infestations) | 0 | 0 | 1
Otitis media (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 2 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 2
Tinea cruris (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 7 | 5 | 5
Urinary tract infection (Infections and infestations) | 1 | 1 | 2
Viral pharyngitis (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 1
Animal scratch (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 2 | 3
Excoriation (Injury, poisoning and procedural complications) | 1 | 1 | 2
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 2 | 0
Heat stroke (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 2 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 4 | 3
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 1 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Postoperative fever (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 2 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 4 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 3 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 2
Blood cholesterol increased (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 1 | 1 | 4
Blood prolactin increased (Investigations) | 2 | 4 | 4
Blood triglycerides increased (Investigations) | 0 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 1
Glucose urine present (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 1 | 1 | 1
Neutrophil count decreased (Investigations) | 1 | 0 | 0
Occult blood (Investigations) | 0 | 0 | 1
Protein urine present (Investigations) | 0 | 1 | 1
Urine ketone body present (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 2 | 3
Weight increased (Investigations) | 3 | 1 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 7 | 2 | 7
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 4 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 5 | 2
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ageusia (Nervous system disorders) | 1 | 0 | 0
Akathisia (Nervous system disorders) | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 1 | 0
Coordination abnormal (Nervous system disorders) | 1 | 1 | 0
Crying (Nervous system disorders) | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 9 | 21 | 19
Dizziness postural (Nervous system disorders) | 3 | 3 | 2
Dysgeusia (Nervous system disorders) | 3 | 0 | 4
Headache (Nervous system disorders) | 25 | 23 | 28
Hyperkinesia (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 3 | 2 | 3
Hypogeusia (Nervous system disorders) | 0 | 1 | 1
Lethargy (Nervous system disorders) | 1 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 2 | 2 | 0
Migraine (Nervous system disorders) | 1 | 1 | 2
Paraesthesia (Nervous system disorders) | 3 | 0 | 1
Parosmia (Nervous system disorders) | 1 | 0 | 1
Poor quality sleep (Nervous system disorders) | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 0
Sedation (Nervous system disorders) | 2 | 1 | 2
Somnolence (Nervous system disorders) | 12 | 12 | 15
Speech disorder (Nervous system disorders) | 1 | 0 | 2
Syncope (Nervous system disorders) | 1 | 0 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 2
Tongue paralysis (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 2 | 2 | 4
Abnormal dreams (Psychiatric disorders) | 10 | 9 | 12
Agitation (Psychiatric disorders) | 0 | 2 | 1
Alcoholic hangover (Psychiatric disorders) | 1 | 0 | 0
Anger (Psychiatric disorders) | 1 | 1 | 1
Anorgasmia (Psychiatric disorders) | 1 | 1 | 4
Anxiety (Psychiatric disorders) | 4 | 5 | 4
Bipolar I disorder (Psychiatric disorders) | 0 | 1 | 0
Bruxism (Psychiatric disorders) | 2 | 0 | 2
Confusional state (Psychiatric disorders) | 1 | 1 | 0
Depression (Psychiatric disorders) | 9 | 5 | 4
Derealisation (Psychiatric disorders) | 2 | 1 | 2
Dissociation (Psychiatric disorders) | 1 | 0 | 2
Eating disorder (Psychiatric disorders) | 1 | 0 | 0
Elevated mood (Psychiatric disorders) | 0 | 1 | 1
Emotional disorder (Psychiatric disorders) | 0 | 0 | 1
Euphoric mood (Psychiatric disorders) | 0 | 0 | 1
Initial insomnia (Psychiatric disorders) | 1 | 2 | 0
Insomnia (Psychiatric disorders) | 10 | 10 | 12
Intentional self-injury (Psychiatric disorders) | 0 | 0 | 1
Libido decreased (Psychiatric disorders) | 3 | 2 | 11
Libido increased (Psychiatric disorders) | 1 | 0 | 0
Loss of libido (Psychiatric disorders) | 0 | 1 | 1
Middle insomnia (Psychiatric disorders) | 1 | 1 | 2
Mood altered (Psychiatric disorders) | 0 | 1 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 1
Nightmare (Psychiatric disorders) | 1 | 0 | 6
Orgasm abnormal (Psychiatric disorders) | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1 | 1
Restlessness (Psychiatric disorders) | 1 | 0 | 3
Self injurious behaviour (Psychiatric disorders) | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0
Sleep inertia (Psychiatric disorders) | 0 | 0 | 2
Suicidal ideation (Psychiatric disorders) | 7 | 9 | 4
Tension (Psychiatric disorders) | 0 | 0 | 1
Terminal insomnia (Psychiatric disorders) | 0 | 0 | 1
Withdrawal syndrome (Psychiatric disorders) | 3 | 5 | 12
Calculus ureteri (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 1
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 4
Polyuria (Renal and urinary disorders) | 0 | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 1
Ejaculation delayed (Reproductive system and breast disorders) | 0 | 2 | 1
Ejaculation disorder (Reproductive system and breast disorders) | 0 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 2 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0 | 0
Premenstrual syndrome (Reproductive system and breast disorders) | 1 | 0 | 0
Sexual dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 4
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Yawning (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Dyshidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6 | 1 | 8
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 3 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 3 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 1 | 0
Hot flush (Vascular disorders) | 5 | 2 | 5
Hypertension (Vascular disorders) | 2 | 0 | 3
Hypotension (Vascular disorders) | 0 | 0 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 2 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0
Spider vein (Vascular disorders) | 0 | 1 | 0
Vasodilatation (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.